CLINICAL TRIAL: NCT05407194
Title: Additional Effect of Collagen/Vitamin C in Exercise Treatment for Patellar Tendinopathy (Jumper's Knee); a Randomized Controlled Trial
Brief Title: Effect of Collagen/Vitamin C in Jumper's Knee; a RCT
Acronym: Jumpfood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gelderse Vallei Hospital (Other)
Responsible Party: Principal Investigator, Rieneke Terink, Scientific researcher, Gelderse Vallei Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL79100.081.21
Record Dates: First submitted 2022-01-08; First posted 2022-06-07 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Patellar Tendinopathy
Keywords: collagen; progressive tendon loading therapy; gelatin; RCT
MeSH Terms: interventions — Collagen; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Investigator
Masking Description: Supplement and placebo will be blinded for participants and researchers working on the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement + progressive tendon loading therapy (Experimental): The intervention consists of a nutritional supplement with 10g hydrolysed collagen and 40 mg vitamin C, in comparison to a placebo supplement consisting of maltodextrin. All participants in both groups will receive education, load management advices and a criteria-based PTLE consisting of 4 stages within the limits of pain during 24-weeks. This (training) intervention has recently been proven to be superior to eccentric training. Participants will be randomly assigned to receive either the nutritional supplement collagen/vitamin C (intervention) or a placebo supplement.
  Interventions: Dietary Supplement: Collagen + vitamin C
- Placebo + progressive tendon loading therapy (Placebo Comparator): The placebo consists of maltodextrin. In comparison the intervention consists of a nutritional supplement with 10g hydrolysed collagen and 40 mg vitamin C. All participants in both groups will receive education, load management advices and a criteria-based PTLE consisting of 4 stages within the limits of pain during 24-weeks. This (training) intervention has recently been proven to be superior to eccentric training. Participants will be randomly assigned to receive either the nutritional supplement collagen/vitamin C (intervention) or a placebo supplement.
  Interventions: Dietary Supplement: Collagen + vitamin C

INTERVENTIONS:
Dietary Supplement: Collagen + vitamin C — Participants take the supplement (or placebo) every day for 24 weeks. On three days per week they perform tendon loading exercises.

SUMMARY:
Patellar tendinopathy (PT) is a tendon overuse injury with high prevalence rates in elite and recreational athletes. PT sometimes results in a prolonged absence from sport participation, hampering individuals to achieve their desired performance levels and to benefit from the health related effects of sports participation. Many treatment options are used but management of PT remains challenging. Current treatment involves progressive education, load management and tendon loading exercises (PTLE). Recent studies have shown that nutrition can positively affect collagen synthesis in musculoskeletal tissues. A study showed that supplementing 15g of gelatine combined with 50mg of Vitamin C, 1 hour before loading exercises, resulted in an increase in whole body collagen synthesis and increased mechanics and collagen content of human engineered ligaments. However the effectiveness of oral supplementation of hydrolysed collagen in combination with vitamin C in athletes with PT has not been studied in a randomized controlled trial yet.

Objective: The primary aim of this RCT is to evaluate whether the use of oral supplementation of hydrolysed collagen/vitamin C in addition to usual care (education, load management and PTLE) is superior to usual care and placebo on VISA-P score after 12, 24 and 52 weeks for athletes with PT. The secondary aim of this RCT is to evaluate whether the use of oral supplementation of hydrolysed collagen/vitamin C in addition to usual care (education, load management and PTLE) is superior to usual care and placebo on other clinical outcome parameters, functional tests and tendon structure after 12 and 24 weeks for athletes with PT.

DETAILED DESCRIPTION:
Rationale: Patellar tendinopathy (PT) is a tendon overuse injury with high prevalence rates in elite and recreational athletes. PT sometimes results in a prolonged absence from sport participation, hampering individuals to achieve their desired performance levels and to benefit from the health related effects of sports participation. Many treatment options are used but management of PT remains challenging. Current treatment involves progressive education, load management and tendon loading exercises (PTLE). Recent studies have shown that nutrition can positively affect collagen synthesis in musculoskeletal tissues. A study showed that supplementing 15g of gelatine combined with 50mg of Vitamin C, 1 hour before loading exercises, resulted in an increase in whole body collagen synthesis and increased mechanics and collagen content of human engineered ligaments. However the effectiveness of oral supplementation of hydrolysed collagen in combination with vitamin C in athletes with PT has not been studied in a randomized controlled trial yet.

Objective: The primary aim of this RCT is to evaluate whether the use of oral supplementation of hydrolysed collagen/vitamin C in addition to usual care (education, load management and PTLE) is superior to usual care and placebo on VISA-P score after 12, 24 and 52 weeks for athletes with PT. The secondary aim of this RCT is to evaluate whether the use of oral supplementation of hydrolysed collagen/vitamin C in addition to usual care (education, load management and PTLE) is superior to usual care and placebo on other clinical outcome parameters, functional tests and tendon structure after 12 and 24 weeks for athletes with PT.

Study design: The JUMPFOOD-study is a double blinded, 2-armed randomized placebo controlled trial which investigates the effectiveness of oral supplementation of hydrolysed collagen and vitamin C combined with progressive tendon loading exercise compared to only progressive tendon loading exercises in athletes with PT.

Study population: Recreational, competitive and professional male and female athletes from different kinds of sports will be included. Inclusion criteria: age 16-40 years old; history of focal knee pain for at least 12 weeks localized in the region of the patellar tendon in association with training and competition; playing sports for at least once a week for at least one year; palpation tenderness to the corresponding painful area on the patellar tendon; Victorian Institute of Sports Assessment - Patella (VISA-P) score < 80 out of 100 points.

Intervention: The intervention consists of a nutritional supplement with 10g hydrolysed collagen and 40 mg vitamin C, in comparison to a placebo supplement consisting of maltodextrin. All participants in both groups will receive education, load management advices and a criteria-based PTLE consisting of 4 stages within the limits of pain during 24-weeks. This (training) intervention has recently been proven to be superior to eccentric training. Participants will be randomly assigned to receive either the nutritional supplement collagen/vitamin C (intervention) or a placebo supplement.

Main study parameters/endpoints: The primary outcome measure will be the change in the Dutch version of the VISA-P score. This simple, validated, reliable and injury-specific questionnaire scores the severity of patellar tendinopathy and is sensitive to small changes in symptoms. It was specifically designed for patellar tendinopathy, rating pain, symptoms, simple test of function and the ability to participate in tendon-loading sports [1]. A VISA-P score of 100 indicates no pain, maximum function and maximum ability to play sports. The score decreases with increasing severity of symptoms of PT. The VISA-P questionnaire will be self-administered at baseline, and after 6, 12, 18, 24 and 52 weeks follow-up. Secondary outcomes will include: Pain during functional tests, advanced imaging methods and tendon structure and stiffness measurements (MRI, ultrasound, UTC, Myoton), blood levels of amino acids and inflammatory markers measured in blood, and dietary habits, that will all be measured at baseline, at 12 weeks and at 24 weeks of follow-up. In addition, data on the compliance with the exercise program and supplement intake, training and competition load will be collected weekly using an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 - 40 years old (the chosen age range will minimize chances of other conditions causing anterior knee pain such as osteoarthritis among patients above 40 years and osteochondrotic diseases like Sinding-Larsen-Johansson syndrome and Osgood-Schlatter disease among patients below the age of 16).
* History of focal knee pain in patellar tendon or its patellar or tibial insertion in association with training and/or competition.
* Current symptom duration of at least 12 weeks.
* Sports participation at least once a week for at least one year.
* Palpation tenderness to the corresponding painful area on the patellar tendon.
* Focal patellar tendon pain during patellar tendon loading with a pain provocation test (single leg decline squat and/or single leg jump squat)
* Victorian Institute of Sports Assessment (VISA-P) score < 80 out of 100 points.
* Willingness to take (non-vegetarian) nutritional supplements.

Exclusion Criteria:

* Known presence of inflammatory joint diseases (e.g. spondylarthropathy, gout or rheumatoid arthritis) or familial hypercholesterolaemia.
* Daily use of drugs with a putative effect on the patellar tendon in the preceding year (e.g. fluoroquinolones and statins)
* Knee surgery without a full completion of the rehabilitation program in the history of the index knee
* Previous patellar tendon rupture of the index knee
* Local injection therapy with corticosteroids, other drugs, blood, platelet rich plasma or stem cells in the preceding 12 months
* Acute knee injuries, including patellar tendon injuries with an acute onset
* Inability to perform the PTLE program
* Participation in other concomitant treatment programs
* Signs or symptoms of other coexisting knee pathology on physical examination (such as patellofemoral pain syndrome, joint effusion and joint line tenderness) or additional diagnostics when found necessary by the sports physician (Chondral lesion of the patella or trochlea on MRI or prepatellar bursitis on US).
* Already using collagen supplementation
* Giving blood donation in a period of two months prior to each test day
* Being pregnant or wish to become pregnant in the upcoming year
* Abuse of hard drugs
* An alcohol consumption >21 units/week (men) or >14 units/week (women)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
VISA-P Score | after 6 weeks follow-up
  The primary outcome measure will be the change in the Dutch version of the VISA-P score. This simple, validated, reliable and injury-specific questionnaire scores the severity of patellar tendinopathy and is sensitive to small changes in symptoms. It was specifically designed for patellar tendinopathy, rating pain, symptoms, simple test of function and the ability to participate in tendon-loading sports [1]. A VISA-P score of 100 indicates no pain, maximum function and maximum ability to play sports. The score decreases with increasing severity of symptoms of PT. The VISA-P questionnaire will be self-administered at baseline, and after 6, 12, 18, 24 and 52 weeks follow-up
VISA-P Score | after 12 weeks follow-up
  The primary outcome measure will be the change in the Dutch version of the VISA-P score. This simple, validated, reliable and injury-specific questionnaire scores the severity of patellar tendinopathy and is sensitive to small changes in symptoms. It was specifically designed for patellar tendinopathy, rating pain, symptoms, simple test of function and the ability to participate in tendon-loading sports [1]. A VISA-P score of 100 indicates no pain, maximum function and maximum ability to play sports. The score decreases with increasing severity of symptoms of PT. The VISA-P questionnaire will be self-administered at baseline, and after 6, 12, 18, 24 and 52 weeks follow-up
VISA-P Score | after 18 weeks follow-up
  The primary outcome measure will be the change in the Dutch version of the VISA-P score. This simple, validated, reliable and injury-specific questionnaire scores the severity of patellar tendinopathy and is sensitive to small changes in symptoms. It was specifically designed for patellar tendinopathy, rating pain, symptoms, simple test of function and the ability to participate in tendon-loading sports [1]. A VISA-P score of 100 indicates no pain, maximum function and maximum ability to play sports. The score decreases with increasing severity of symptoms of PT. The VISA-P questionnaire will be self-administered at baseline, and after 6, 12, 18, 24 and 52 weeks follow-up
VISA-P Score | after 24 weeks follow-up
  The primary outcome measure will be the change in the Dutch version of the VISA-P score. This simple, validated, reliable and injury-specific questionnaire scores the severity of patellar tendinopathy and is sensitive to small changes in symptoms. It was specifically designed for patellar tendinopathy, rating pain, symptoms, simple test of function and the ability to participate in tendon-loading sports [1]. A VISA-P score of 100 indicates no pain, maximum function and maximum ability to play sports. The score decreases with increasing severity of symptoms of PT. The VISA-P questionnaire will be self-administered at baseline, and after 6, 12, 18, 24 and 52 weeks follow-up
VISA-P Score | after 52 weeks follow-up
  The primary outcome measure will be the change in the Dutch version of the VISA-P score. This simple, validated, reliable and injury-specific questionnaire scores the severity of patellar tendinopathy and is sensitive to small changes in symptoms. It was specifically designed for patellar tendinopathy, rating pain, symptoms, simple test of function and the ability to participate in tendon-loading sports [1]. A VISA-P score of 100 indicates no pain, maximum function and maximum ability to play sports. The score decreases with increasing severity of symptoms of PT. The VISA-P questionnaire will be self-administered at baseline, and after 6, 12, 18, 24 and 52 weeks follow-up

SECONDARY OUTCOMES:
Pain during functional tests | after 12 weeks follow-up
  During several functional tests, pain will be measured on a visual analogue scale, with 0 meaning no pain and 10 meaning unbearable pain, at baseline, 12 weeks and 24 weeks of follow-up.
Pain during functional tests | after 24 weeks follow-up
  During several functional tests, pain will be measured on a visual analogue scale, with 0 meaning no pain and 10 meaning unbearable pain, at baseline, 12 weeks and 24 weeks of follow-up.
Imaging methods | after 12 weeks follow-up
  Several imaging methods will be performed to identify the physiological parameter tendon structure shown in percentages healthy and damaged cells, at baseline, 12 weeks and 24 weeks of follow-up.
Imaging methods | after 24 weeks follow-up
  Several imaging methods will be performed to identify the physiological parameter tendon structure shown in percentages healthy and damaged cells, at baseline, 12 weeks and 24 weeks of follow-up.
Stiffness measurement | after 12 weeks follow-up
  The physiological parameter stiffness of the tendon will be measured in N/m, at baseline, 12 weeks and 24 weeks of follow-up.
Stiffness measurement | after 24 weeks follow-up
  The physiological parameter stiffness of the tendon will be measured in N/m, at baseline, 12 weeks and 24 weeks of follow-up.
Blood levels of amino acids | after 12 weeks follow-up
  Concentration of amino acids in blood will be measured at baseline, 12 weeks and after 24 weeks of follow-up
Blood levels of amino acids | after 24 weeks follow-up
  Concentration of amino acids in blood will be measured at baseline, 12 weeks and after 24 weeks of follow-up
Blood levels of inflammatory markers | after 12 weeks follow-up
  Concentration in blood of the inflammatory markers BSE and CRP will be measured at baseline, 12 weeks and after 24 weeks of follow-up
Blood levels of inflammatory markers | after 24 weeks follow-up
  Concentration in blood of the inflammatory markers BSE and CRP will be measured at baseline, 12 weeks and after 24 weeks of follow-up
Dietary habits | baseline
  Dietary habits (nutritional intake) will be measured at the start and end of the intervention period using a diary.
Dietary habits | after 24 weeks
  Dietary habits (nutritional intake) will be measured at the start and end of the intervention period using a diary.
Compliance | Weekly during the intervention, up to 24 weeks follow-up
  Data on the compliance with the exercise program and supplement intake, but also on training and competition load will be collected weekly using an online questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gelderse Vallei Hospital, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
patient data, not able to share

REFERENCES:
- [Derived] van Dam L, Terink R, Mensink M, de Vos RJ, Zwerver J. The JUMPFOOD study: additional effect of hydrolyzed collagen and vitamin C to exercise treatment for patellar tendinopathy (jumper's knee) in athletes-study protocol for a double-blind randomized controlled trial. Trials. 2023 Nov 28;24(1):768. doi: 10.1186/s13063-023-07783-2. PMID 38017500